CLINICAL TRIAL: NCT05170581
Title: Efficacy and Safety of Sintilimab Combined With Platinum-containing Chemotherapy in Neoadjuvant Treatment of Resectable Stage ⅡB～ⅢA Non-small Cell Lung Cancer
Brief Title: Clinical Study of Sintilimab Combined With Chemotherapy in Neoadjuvant Treatment of Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-003
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Sintilimab; Neoadjuvant Treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 inhibitor combined with chemotherapy (Experimental): Sintilimab will be administered one day before platinum-containing chemotherapy.
  Interventions: Drug: Sintilimab Combined with Platinum-containing Chemotherapy

INTERVENTIONS:
Drug: Sintilimab Combined with Platinum-containing Chemotherapy — Admininster Sintilimab and platinum-containing chemotherapy in neoadjuvant treatment of resectable stage ⅡB～ⅢA Non-small Cell Lung Cancer
  Other Names: PD-1 inhibitor combined with chemotherapy

SUMMARY:
By exploring the feasibility, effectiveness and safety of neoadjuvant therapy with Sintilimab combined with platinum-containing chemotherapy in patients with resectable Stage ⅡB-ⅢA NSCLC, we will provide new treatment options and strategies for stage ⅡB-ⅢA NSCLC.

DETAILED DESCRIPTION:
The distant recurrence rate after radical surgery for early and partial locally advanced NSCLC is high, while the benefit degree of neoadjuvant chemotherapy is not satisfactory. The purpose of this study is to explore the feasibility, effectiveness and safety of neoadjuvant therapy with Sintilimab combined with platinum-containing chemotherapy in patients with resectable Stage ⅡB-ⅢA NSCLC.

In addition to exploring the advantages of clinical efficacy of combination therapy, the analysis of biomolecular markers will be used to further understand the effects of combination therapy mode on immune activation and tumor immune microenvironment, and to explore potential biomarkers for predicting treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent prior to implementing any trial-related procedures; 2. Male or female ≥18 years old and ≤75 years old; 3. Cytological or histological diagnosis of non-small cell lung cancer; 4. According to the efficacy evaluation criteria for solid tumors (RECIST version 1.1), at least one lesion can be measured on imaging; 5. Untreated stage ⅰ B - ⅲ A non-small cell lung cancer (TNM staging according to UICC/AJCC Edition 8); 6. Primary tumor can be biopsied; 7. Patients who agree to receive radical surgical treatment; 8. Patients who can be resected by surgeons and have no contraindications; 9. ECOG score 0-1; 10. Expected survival time > 6 months; 11. Adequate organ function, subject will meet the following laboratory criteria: 1) Absolute value of neutrophils (ANC) ≥1.5x10^9/L without the use of granulocyte colony-stimulating factor in the last 14 days. 2) Platelets ≥100×10^9/L in the last 14 days without blood transfusion. 3) In the absence of blood transfusion or erythropoietin in the last 14 days, hemoglobin>9 g/dL. 4) Total bilirubin ≤1.5× upper normal value (ULN); 5) Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN 6) Serum creatinine ≤1.5×ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥60 mL /min; 7) Good coagulation function, defined as international standardized ratio (INR) or prothrombin time (PT) ≤1.5 ULN; 8) Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range may be enrolled; 9) The myocardial enzyme profile is within the normal range (if the investigator comprehensively determines that the simple laboratory abnormality is not clinically significant, it is allowed to be included in the group); 12. For female subjects of reproductive age, a negative urine or serum pregnancy test should be performed within 3 days prior to receiving the first study drug administration (day 1 of cycle 1). If a urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is requested. Women of childbearing age were defined as at least 1 year after menopause or having undergone surgical sterilization or hysterectomy; If there is a risk of pregnancy, all subjects (both men and women) are required to use a contraceptive with an annual failure rate of less than 1% for the entire treatment period up to 120 days after the last study drug (or 180 days after the last chemotherapeutic drug).

Exclusion Criteria:

1. Malignant diseases other than NSCLC were diagnosed within 5 years prior to first administration (excluding radical basal cell carcinoma of the skin, squamous carcinoma of the skin, and/or radical resected carcinoma in situ); 2. Are currently participating in an interventional clinical study or have been treated with another study drug or study device within 4 weeks prior to initial administration; 3. Prior treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs that target another stimulating or co-inhibiting T-cell receptor (e.g., CTLA-4, OX-40, CD137); 4. Received systemic systemic therapy with anti-tumor indications of Proprietary Chinese medicines or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local use to control pleural effusion) within 2 weeks before the first administration; 5. An active autoimmune disease requiring systemic therapy (e.g., palliative drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years prior to first dosing. Alternative therapies (e.g. thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary dysfunction) are not considered systemic; 6. Were receiving systemic glucocorticoid therapy (excluding nasal spray, inhalation, or other topical glucocorticoid) or any other form of immunosuppressive therapy within 7 days prior to initial dosing; Note: Physiological doses of glucocorticoids (≤10 mg/ day of prednisone or equivalent) are permitted; 7. Allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation is known; 8. Those who are known to be allergic to the active ingredient or excipient of sindilizumab; 9. Has not fully recovered from toxicity and/or complications associated with any intervention prior to initiation of treatment (i.e., ≤ grade 1 or baseline, excluding fatigue or hair loss); 10. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive); 11. Untreated active hepatitis B (defined as HBsAg positive with hbV-DNA copy number greater than the upper limit of the normal value in the laboratory department of the research center); Note: Hepatitis B subjects who meet the following criteria can also be enrolled: 1) HBV viral load before initial administration < 1000 copies/mL (200 IU/ml). Subjects should receive anti-HBV therapy throughout study chemotherapy to avoid virus reactivation 2) For subjects resistant to HBc (+), HBsAg (-), anti-HBS (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of virus reactivation is required 12. Active HCV-infected subjects (HCV antibody positive and HCV-RNA level above the detection limit); 13. Received live vaccine within 30 days prior to initial administration (cycle 1, day 1); Note: Acceptance of injectable inactivated virus vaccine against seasonal influenza is permitted within 30 days prior to first administration; Intranasally administered live attenuated flu vaccines are not allowed. 14. Pregnant or lactating women; 15. Presence of any serious or uncontrollable systemic illness, such as: 1) Serious and uncontrollable abnormalities in the rhythm, conduction or morphology of resting electrocardiogram, such as complete left bundle branch block, heart block above degree ⅱ, ventricular arrhythmia or atrial fibrillation; 2) Unstable angina pectoris, congestive heart failure, NYHA grade ≥ 2 chronic heart failure; 3) Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months prior to treatment inclusion; 4) Poor blood pressure control (systolic > 140 mmHg, diastolic > 90 mmHg); 5) A history of non-infectious pneumonia requiring glucocorticoid treatment within 1 year prior to initial administration, or the current presence of clinically active interstitial lung disease; 6) Active tuberculosis; 7) The presence of active or uncontrolled infections requiring systemic treatment; 8) Clinical active diverticulitis, abdominal abscess and gastrointestinal obstruction; 9) Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis; 10) Poor control of diabetes (FBG > 10mmol/L); 11) Urine routine showed urine protein ≥++, and confirmed 24-hour urine protein quantity > 1.0g; 12) Patients with mental disorders and unable to cooperate with treatment; Any medical history or disease evidence that may interfere with the study results, prevent the subjects from participating fully in the study, abnormal values of treatment or laboratory tests, or other conditions that the investigator considers inappropriate for the study because of other potential risks that the investigator considers inappropriate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Major pathological remission | 3 years
  Residual tumor cells were less than 10% in postoperative specimen pathology
Event-free survival | 3 years
  The time from enrollment to occurrence of any event, including death, disease progression, change of chemotherapy regimen, change to chemotherapy, addition of other treatments, occurrence of fatal or intolerable side effects.

SECONDARY OUTCOMES:
Pathological complete remission | 3 years
  No tumor cells were found in postoperative specimen pathology
Overall Survival | 3 years
  Time from randomization to death (from any cause)
Disease-free survival | 3 years
  The time between randomization and relapse of disease or death (from any cause)
Objective remission rate | 3 years
  The proportion of patients whose tumor volume shrinks to a predetermined value and maintains the minimum time limit is the sum of complete and partial responses.

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Liu, Principal Investigator — The Second Affiliated Hospital of Shandong First Medical Universuty
Locations (1):
- The Second Affiliated Hospital of Shandong First Medical University, Tai’an, Shandong, China

REFERENCES:
- [Background] Provencio M, Nadal E, Insa A, Garcia-Campelo MR, Casal-Rubio J, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Pereira E, Royuela A, Casarrubios M, Salas Anton C, Parra ER, Wistuba I, Calvo V, Laza-Briviesca R, Romero A, Massuti B, Cruz-Bermudez A. Neoadjuvant chemotherapy and nivolumab in resectable non-small-cell lung cancer (NADIM): an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Nov;21(11):1413-1422. doi: 10.1016/S1470-2045(20)30453-8. Epub 2020 Sep 24. PMID 32979984
- [Background] Gao S, Li N, Gao S, Xue Q, Ying J, Wang S, Tao X, Zhao J, Mao Y, Wang B, Shao K, Lei W, Wang D, Lv F, Zhao L, Zhang F, Zhao Z, Su K, Tan F, Gao Y, Sun N, Wu D, Yu Y, Ling Y, Wang Z, Duan C, Tang W, Zhang L, He S, Wu N, Wang J, He J. Neoadjuvant PD-1 inhibitor (Sintilimab) in NSCLC. J Thorac Oncol. 2020 May;15(5):816-826. doi: 10.1016/j.jtho.2020.01.017. Epub 2020 Feb 6. PMID 32036071